CLINICAL TRIAL: NCT04067635
Title: Primary Mitral Regurgitation Reverse Remodeling
Brief Title: Primary Mitral Regurgitation Repair
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Eric Y. Yang, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Eric Y. Yang, MD PhD, Principal Investigator, Houston Methodist Hospital Physician, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Other Study IDs: Pro00018490
Record Dates: First submitted 2019-08-21; First posted 2019-08-26 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Mitral Valve Insufficiency; Mitral Valve Prolapse; Chronic Mitral Disease; Mitral Regurgitation; Mitral Valve Disease; Degenerative Mitral Valve Disease; Myxomatous Mitral Valve Degeneration; Ventricular Remodeling
Keywords: Mitral Valve Annuloplasty; Mitral Regurgitation; Primary Mitral Regurgitation; Chronic Mitral Regurgitation; Ventricular Reverse Remodeling; Ventricular Recovery
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Prolapse; Ventricular Remodeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole Blood, Serum, Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Conservative Arm: Participants are followed by the research team conservatively. Participants in this arm may choose to undergo any valvular intervention at the discretion of their treating clinical team.
- Surgical Arm: Participants have already elected upfront to undergo surgical repair (at least, mitral annuloplasty) with their treating clinical team, just prior to enrollment into this study.

SUMMARY:
This longitudinal cohort study evaluates the relationship of myocardial tissue markers characteristics assessed by cardiac MRI, with clinical measures of symptoms and functions in adults with primary mitral regurgitation. Participants are followed conservatively or may choose to undergo surgical repair at the discretion of their clinical team.

DETAILED DESCRIPTION:
The transition from compensated to decompensated chronic primary mitral regurgitation remains poorly understood in the clinical setting. Changes at the myocardial tissue level, such as scar formation and decreased contractility, have been implicated in the end stage, decompensated phase of this disease entity.

Advances in cardiac MRI (CMR) have enabled non-invasive characterization of the myocardial tissue components, such as cardiomyocyte volume and extracellular matrix, and tissue contractility. These measures have been well validated in various cardiac pathologies with biopsy studies but only at single time points.

In this study, adults with isolated chronic primary regurgitation will be followed conservatively over at least a year to determine the natural progression of these CMR-derived markers over time and to investigate the prognostic potential of these markers for clinically assessed functional capacity and symptoms. These participants may elect to undergo any valvular intervention at the discretion of their treating clinical team.

Alongside this arm, similar adults with isolated chronic primary regurgitation will be recruited, who have elected upfront to undergo surgical repair. These patients will be similarly studied to determine reverse remodeling of these CMR-derived markers over time and to investigate the prognostic potential of these markers for the same clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Isolated mitral regurgitation

   1. of any primary mechanism and
   2. of moderate-to-severe (Sellers 3+) or greater severity, assessed by any imaging modality (echocardiography, angiography, cardiac MRI)
3. Able to receive gadolinium-based contrast agent (estimated glomerular filtration rate >30 mL/min/1.73 m2, no prior allergy to gadolinium contrast agents)

Exclusion Criteria:

1. Refusal to consent
2. Pregnancy during the study
3. Hemodynamically or clinically unstable
4. Inability to undergo a CMR scan, which can include the following reasons: severe claustrophobia, ferromagnetic implants, implanted defibrillator, pacemaker, or abandoned pacemaker leads, cochlear implants, unable to lie flat
5. Other diseases known to influence myocardial fibrosis development (coronary artery disease, diabetes mellitus, uncontrolled hypertension, infiltrative cardiomyopathy, myocarditis, hypertrophic cardiomyopathy, any cardiac tumors, moderate or more valvular heart disease other than primary mitral valve regurgitation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cardiac MRI referral base, valve specialty clinic
Sampling Method: Non-Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2018-05-25 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Changes in cardiomyopathy symptom score | Baseline, 6 (+/-3) months, >12 months
  Heart failure symptom scores will be tracked to monitor for changes in symptom burden at 2 subsequent timepoints. Scores are derived from a validated cardiomyopathy symptom patient-reported outcome measure instrument. The full name of the instrument is the Kansas City Cardiomyopathy Questionnaire Short Form (aka KCCQ-12) licensed by CV Outcomes, Inc. Only a complete score is recorded. The full range of scores scale from 0 to 100, with higher scores indicating lower symptom burden.
Changes in distance measured on 6-Minute Walk Test | Baseline, 6 (+/-3) months, >12 months
  Distance (meters) walked using a standardized 6-minute walk protocol will be tracked to monitor for changes in functional capacity at 2 subsequent timepoints.

SECONDARY OUTCOMES:
Late gadolinium myocardial enhancement | Baseline, 6 (+/-3) months, >12 months
  Semi-quantitative measure of left ventricular replacement fibrosis burden using cardiac MRI techniques with gadolinium-based contrast agents. The quantity measured is the percentage of left ventricular myocardial volume found to have late gadolinium enhancement.
Myocardial extracellular volume fraction | Baseline, 6 (+/-3) months, >12 months
  Extracellular volume fraction measure derived using T1 mapping from cardiac MRI techniques. The quantity measured is the proportion of extracellular matrix volume to cardiomyocyte volume.
Cardiac Morphology | Baseline, 6 (+/-3) months, >12 months
  Cardiac MRI measures from cine images of cardiac chamber dimensions (milliliters) at end-diastolic and end-systolic cardiac phases.
Cardiovascular Flow Volumes | Baseline, 6 (+/-3) months, >12 months
  Cardiovascular MRI measures from phase contrast cine images of flow (mL/s) through major vessels. The flow quantity is integrated over a cardiac cycle to produce a volume (mL) per beat.
Ventricular Mass | Baseline, 6 (+/-3) months, >12 months
  Cardiac MRI measures of left ventricular myocardial mass (grams)

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States